CLINICAL TRIAL: NCT03768024
Title: A Single-Dose, Randomized, Double Blind, Placebo and Active Controlled Cross-Over Study to Evaluate the Abuse Potential of Three Doses of GRT0151Y in Adult Non-dependent Recreational Opiate Users
Brief Title: A Clinical Study in Healthy Adults Who Sometimes Take Drugs for Pleasure Which Aims to Evaluate Whether GRT0151Y is Likely to be Abused
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP0151Y/13; PK877A (Other: Sponsor)
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Pain; Acute Pain
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Intervention Model Description: Qualified participants for the treatment phase will be randomized to 1 of 7 treatment-sequences based on a computer generated randomization schedule. Participants will receive all 7 treatments in the order specified by the treatment sequence according to a 7-sequence, 7-period balanced design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Treatment A: GRT0151Y 100 mg (Experimental): Treatment A: GRT0151Y 100 mg free base: 2 × GRT0151Y 50 mg capsules and 6 placebo capsules. A single dose comprised 8 capsules in total which will be taken with water and in a fasted state.
  Interventions: Drug: GRT0151Y 50 mg capsule; Drug: Matching placebo
- Treatment B: GRT0151Y 200 mg (Experimental): Treatment B: GRT0151Y 200 mg free base: 4 × GRT0151Y 50 mg capsules and 4 placebo capsules. A single dose comprised 8 capsules in total which will be taken with water and in a fasted state.
  Interventions: Drug: GRT0151Y 50 mg capsule; Drug: Matching placebo
- Treatment C: GRT0151Y 400 mg (Experimental): Treatment C: GRT0151Y 400 mg free base: 8 × GRT0151Y 50 mg capsules. A single dose comprised 8 capsules in total which will be taken with water and in a fasted state.
  Interventions: Drug: GRT0151Y 50 mg capsule
- Treatment D: Matching placebo (Experimental): Treatment D: Matching placebo to GRT0151Y and hydromorphone IR: 8 placebo capsules. A single dose comprised 8 capsules in total which will be taken with water and in a fasted state.
  Interventions: Drug: Matching placebo
- Treatment E: Hydromorphone IR 4 mg (Experimental): Treatment E: Hydromorphone IR 4 mg: 1 × hydromorphone IR 4 mg tablet (encapsulated) and 7 placebo capsules. A single dose comprised 8 capsules in total which will be taken with water and in a fasted state.
  Interventions: Drug: Hydromorphone IR 4 mg; Drug: Matching placebo
- Treatment F: Hydromorphone IR 8 mg (Experimental): Treatment F: Hydromorphone IR 8 mg: 2 × hydromorphone IR 4 mg tablet (encapsulated) and 6 placebo capsules. A single dose comprised 8 capsules in total which will be taken with water and in a fasted state.
  Interventions: Drug: Hydromorphone IR 4 mg; Drug: Matching placebo
- Treatment G: Hydromorphone IR 16 mg (Experimental): Treatment G: Hydromorphone IR 16 mg: 4 × hydromorphone IR 4 mg tablet (encapsulated) and 4 placebo capsules. A single dose comprised 8 capsules in total which will be taken with water and in a fasted state.
  Interventions: Drug: Hydromorphone IR 4 mg; Drug: Matching placebo

INTERVENTIONS:
Drug: GRT0151Y 50 mg capsule — GRT0151Y 50 mg capsule
  Arms: Treatment A: GRT0151Y 100 mg; Treatment B: GRT0151Y 200 mg; Treatment C: GRT0151Y 400 mg
Drug: Hydromorphone IR 4 mg — Hydromorphone IR 4 mg tablet (encapsulated)
  Arms: Treatment E: Hydromorphone IR 4 mg; Treatment F: Hydromorphone IR 8 mg; Treatment G: Hydromorphone IR 16 mg
Drug: Matching placebo — Matching placebo
  Arms: Treatment A: GRT0151Y 100 mg; Treatment B: GRT0151Y 200 mg; Treatment D: Matching placebo; Treatment E: Hydromorphone IR 4 mg; Treatment F: Hydromorphone IR 8 mg; Treatment G: Hydromorphone IR 16 mg

SUMMARY:
The purpose of this clinical study was to evaluate whether healthy adults, who sometimes take drugs for pleasure, are likely to abuse GRT0151Y. This abuse potential is assessed at three different doses of GRT0151Y.

During a Qualification Phase, a single dose of hydromorphone IR 8 mg and a single dose of placebo were separately administered orally over 4 days in a randomized, double-blinded manner.

During the Treatment Phase, single doses of GRT0151Y free base (100 mg, 200 mg and 400 mg), hydromorphone Immediate-release (IR) (4 mg, 8 mg, and 16 mg), and placebo were administered orally over 7 Treatment Periods.

Participants received the treatments according to a 7-sequence, 7-period balanced design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 55 years of age, inclusive.
* Acceptable body mass index (BMI) (weight [kilograms]/height (square meter) range of 19 to 30 kilograms per square meter, inclusive).
* Signed an informed consent document indicating that they understand the purpose of and procedures required for the study, and are willing to participate in the study.
* Participants with a history of recreational opiate use (defined as nontherapeutic use at least 10 times in the past year and at least once in the last 12 weeks prior to enrolment) but not dependent on opiates Diagnostic and Statistical Manual of Mental Disorders-4th edition (DSM-IV criteria).
* Participants must consent to use a medically acceptable method of contraception throughout the entire study period, including washout periods. Men must confirm that, when having sexual intercourse with women of childbearing potential (i.e., women who are not surgically sterilized, or and not at least 2 years post-menopausal), they will use a condom from the time of the first dose until 4 weeks after the last dose and that the respective partner will use an additional contraceptive method. Men may be included if surgically sterile. For females of childbearing potential only: adequate contraception is defined as any form of hormonal contraception or intra-uterine device that needs to be in place for a period of at least two months prior to enrolment. Additional barrier contraception must be used for the duration of the study, defined as the time from the enrolment visit to the final examination, and for at least one full month thereafter. A single barrier method alone or abstinence alone is not acceptable. Women of non-childbearing potential may be included if surgically sterile or postmenopausal for at least two years.
* Female participants of childbearing potential must have a negative pregnancy test (beta-Human chorionic gonadotropin) at the enrolment visit and before receiving study drug for each of the double-blind qualification and treatment periods. For females of childbearing potential, the time between the Enrolment Visit and first receipt of drug will be separated by a minimum of 10 days to ensure accuracy of the pregnancy test.
* Participants with a positive urine drug screen (for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, phencyclidine and opiates) upon presentation for study days will be allowed to continue only if the investigator or designee considers that the presence of the drug will not introduce additional risk factors for the study participant, or interfere with study procedures or data integrity. Positive drug screens for select drugs are to be confirmed using quantitative methods such as Gas Chromatography (GC)/Mass Spectrometry (MS) or equivalent, and the investigator or designee's decision to allow participants to continue will take into account the quantitative levels of drug in the participants' urine. Participants may be rescheduled for another treatment session at the investigator's discretion.
* Deemed healthy on the basis of enrolment visit physical examination, medical history, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters (biochemistry, urinalysis, clotting, blood sedimentation rate [BSR], haematology and hepatitis and human immunodeficiency virus [HIV] virus serology). If the results of the laboratory tests or the urinalysis testing are not within the laboratory's reference ranges, the participant can be included only on condition that the investigator or designee judges that the deviations are not clinically relevant and do not interfere with the study objectives.
* Must have a negative breath alcohol analysis at enrolment. A positive alcohol reading is one that is above the error measurement associated with the breathalyzer. Participants presenting a positive alcohol breath test may be allowed to continue in the study only if the investigator (or designee) considers that the presence of breath alcohol does not suggest problematic alcohol consumption, and will not introduce additional risk factors for the study participant, or interfere with study procedures or data integrity.
* Must pass a qualifying session.
* Ability to speak, read and understand English sufficiently in order to understand the nature of the study, to provide written informed consent and to allow completion of all study assessments.

Exclusion Criteria:

* History of, or current substance dependence (except nicotine and caffeine dependence) as defined by the DSM-IV.
* Participants attempting to discontinue their recreational drug use, or who have been in a drug rehabilitation program in the 12 months prior to enrolment.
* History or risk of seizures (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness).
* Positive HIV type 1/2 antibodies, Hepatitis B surface (HBs) antigen, Hepatitis B core (HBc) antibodies (Immunoglobulin G and Immunoglobulin M), Hepatitis C virus (HCV) antibodies.
* Participants with gastrointestinal disease (e.g., paralytic ileus) or constipation or who have clinically significant gastrointestinal problems, including narrowing (pathologic or iatrogenic) of the gastrointestinal tract, or diseases or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Contraindications listed in the current summary of product characteristics of hydromorphone.
* Participants with a history of, or current Chronic Obstructive Pulmonary Disease, or any other lung disease, (e.g., asthma, sleep apnea) that would cause carbon dioxide (CO2) retention.
* Participants with a history of or current cardiovascular dysfunction including marked repolarization abnormality (e.g., suspicious or definite congenital long QT syndrome, resting pulse rate less than or equal to 45 or greater than or equal to 95 beats per minute, and orthostatic or uncontrolled hypotension or hypertension (systolic blood pressure less than or equal to 100 and greater than or equal to 140 Millimeter mercury (mmHg), diastolic blood pressure less than or equal to 50 and greater than or equal to 95 mmHg), or use of co-medication that is known to influence cardiac repolarization substantially, evaluated at enrolment.
* QT/QTc (Bazett) interval greater than 450 milliseconds (males), greater than 470 milliseconds (females).
* Male participants with hemoglobin less than 125 grams per Liter and female participants with hemoglobin less than 115 grams per Liter.
* Blood donation (more than 150 milliliters) within 3 months before starting this study, i.e. first administration of IMP.
* Known contraindications/hypersensitivity to other opioids, naloxone, benzodiazepines, hydromorphone or definite or suspected allergy or hypersensitivity to drugs having similar mechanism of action as the study drug.
* Pregnant or lactating.
* Participants who have used any prescription medication (except for sex-hormone replacement or birth control medications) including known CYP2D6 inhibitors and substrates which lower the seizure threshold within 14 days prior to the first study drug administration or monoamine-oxidase inhibitors (MAOIs) within 21 days prior to the first study drug administration.
* History or presence of co-medication with tricyclics antidepressants (TCA), selective serotonin re-uptake inhibitors (SSRI), serotonin norepinephrine reuptake inhibitors (SNRI), and antiparkinsonian drugs within 30 day prior to the first study drug administration.
* Participants who plan to take prescription medication, over-the-counter, or Natural Health Products during the study, with the exception of birth control medications, sex-hormone replacement, vitamins/minerals and acetominophen (up to 2 grams per day).
* Participants who have taken a new chemical entity under development within the last 30 days prior to receiving the first dose of IMP or longer, if on the basis of pharmacokinetic/pharmacodynamic characteristics, a possible interaction with study objective cannot be reasonably excluded.
* Not able to abstain from drinking of caffeine containing beverages (tea, coffee, chocolate or cola). Participants not able to refrain from smoking more than 20 cigarettes per day.
* Serum creatinine higher than 1.5 x upper limit of normal range, at enrolment.
* Any documented or suspected DSM-IV psychiatric disorder currently or within the past year, or any prior psychiatric condition that might compromise participant safety by increasing the risk of an untoward effect from the study drugs administered in this study as determined by the investigator's or designee's assessment of the Symptom Checklist 90-R (SCL-90-R) results.
* Participants who, in the investigator's opinion, may not be capable of following the study schedule for any reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2007-06-21 (Actual); Primary Completion 2007-10-25 (Actual); Study Completion 2007-10-25 (Actual)

PRIMARY OUTCOMES:
Overall Drug Liking | at 24 hours post-dose
  100-point bipolar VAS ratings after each investigational medicinal product (IMP) administration in response to the statement "Overall, my liking for this drug is". The 100 mm bipolar VAS is anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), to the left with "strong disliking" (score of 0 mm) and to the right with "strong liking" (score of 100 mm).
Overall Drug Liking | at 48 hours post-dose
  100-point bipolar VAS ratings after each investigational medicinal product (IMP) administration in response to the statement "Overall, my liking for this drug is". The 100 mm bipolar VAS is anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), to the left with "strong disliking" (score of 0 mm) and to the right with "strong liking" (score of 100 mm).
Subjective Drug Value (SDV) | at 24 hours post-dose
  The SDV is a proxy measure of reinforcing efficacy that involves a series of independent, theoretical forced choices between drug administered and different monetary values. Participants were asked to choose between receiving another dose of the same drug or an envelope containing a specified amount of money, but they did not receive drug or money as described.
Subjective Drug Value (SDV) | at 48 hours post-dose
  The SDV is a proxy measure of reinforcing efficacy that involves a series of independent, theoretical forced choices between drug administered and different monetary values. Participants were asked to choose between receiving another dose of the same drug or an envelope containing a specified amount of money, but they did not receive drug or money as described.

SECONDARY OUTCOMES:
Addiction Research Center Inventory (ARCI) | pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hours post-dose
  The ARCI contains 5 scales (49-item), which measure: Euphoria: Morphine-Benzedrine Group, 'MBG' scale. Stimulant-like effects: Amphetamine, 'A' scale and Benzedrine Group, 'BG' scale. Dysphoria: Lysergic Acid Diethylamide, 'LSD' scale. Sedation: Pentobarbital-Chlorpromazine-Alcohol Group, 'PCAG' scale.
  Participants indicate their responses by selecting "False" or "True" with a mouse. One point is given for each response that agrees with the scoring direction on the scale (i.e., True items receive a score of 1 if the answer is "True", False items receive a score of 1 if the answer is "False". No points (0) are given when the answer is opposite to the scoring direction). Higher scores indicated higher effects.
Drug Liking "at this moment" | at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours post-dose
  100-point bipolar visual analog scale (VAS) ratings after each IMP administration in response to the statement "At this moment, my liking for this drug is". The 100 millimeter (mm) bipolar VAS is anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), to the left with "strong disliking" (score of 0 mm) and to the right with "strong liking" (score of 100 mm).
Good Effects | at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours post-dose
  100-point unipolar VAS ratings after each IMP administration in response to the statement "At this moment, I can feel good drug effects". The 100 mm unipolar VAS is anchored to the left with 'definitely not' (score of 0 mm) and to the right with 'definitely so' (score of 100).
Bad Effects | at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours post-dose
  100-point unipolar VAS ratings after each IMP administration in response to the statement "At this moment, I can feel bad drug effects". The 100 mm unipolar VAS is anchored to the left with 'definitely not' (score of 0 mm) and to the right with 'definitely so' (score of 100).
Any Effects | at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours post-dose
  100-point unipolar VAS ratings after each IMP administration in response to the statement "At this moment, I can feel a drug effect". The 100 mm unipolar VAS, is anchored to the left with 'definitely not' (score of 0 mm) and to the right with 'definitely so' (score of 100).
Subject-rated Opiate Agonist Scale (SROAS) | at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours post-dose
  16 VAS items: Nodding, Dry Mouth, Turning of Stomach, Skin Itchy, Relaxed, Coasting, Pleasant Sick, Drive [Energy]' Nervous, Good Mood, High, Sleepy, Drunken, Soapbox [Talkative], Rush, and Friendly. Participants will be asked to respond to the following question: "Indicate how much you feel the following symptom right now." These assessments will be administered as a 0-100 VAS anchored by "Not at all" (0) and "Extremely" (100).
Observer-rated | at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours post-dose
  VAS scales (Scratching, Nervous, Drunken, Talkative, Sleepy). A trained observer will respond to each item following a 5-minute period of observation and indicate how the participant appeared during the period. These assessments will be administered as 0 to 100 VAS anchored by "Definitely not" (0) and "Definitely so" (100).
Take Drug Again | at 12, 24, and 48 hours post-dose
  100-point bipolar VAS ratings after each IMP administration in response to the statement "I would take this drug again". The 100 mm bipolar VAS is anchored in the center with a neutral anchor of "neutral" (score of 50 mm), to the left with "definitely not" (score of 0 mm) and to the right with "definitely so" (score of 100 mm).
Divided Attention test (DA) - Time over the road | pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 32 and 48 hours post-dose
  Manual-tracking test with a simultaneous visual target detection component. Participant is provided with joystick and presented with the image of an airplane and a randomly curving road; participant has to position the airplane over the center of the road while being distracted repeatedly by visual targets they have to respond to. Percentage of time over the road will be recorded.
Divided Attention test (DA) - Response latency | pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 32 and 48 hours post-dose
  Manual-tracking test with a simultaneous visual target detection component. Participant is provided with joystick and presented with the image of an airplane and a randomly curving road; participant has to position the airplane over the center of the road while being distracted repeatedly by visual targets they have to respond to. Response latency of correct responses (milliseconds) will be recorded.
Divided Attention test (DA) - Target hits | pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 32 and 48 hours post-dose
  Manual-tracking test with a simultaneous visual target detection component. Participant is provided with joystick and presented with the image of an airplane and a randomly curving road; participant has to position the airplane over the center of the road while being distracted repeatedly by visual targets they have to respond to. Percentage of target hits will be recorded.
Choice Reaction Time (CRT) | pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 32, and 48 hours post-dose
  Choice reaction time (CRT) is a computerized assessment that trains the participant to respond to stimuli presented on the screen. The task requires the participant to react as soon as a colored key appears in one of up to eight locations. The participant must respond by lifting their finger from the central start button and depressing the corresponding response key as quickly as possible. This is the reaction time (RT). Lower scores indicate better performance.
Pharmacokinetic parameter: AUC0-t | Day 1 pre-dose and 0.75, 1.25, 2.25, 4.25 6.25, 8.25 and 12.25 hours post-dose and on Days 2 and 3 at 24.25, 32.25 and 48.25 hours
  Area under the plasma concentration-time curve from dosing time to the last measured concentration equal or above the lower limit of quantification (LLOQ)
Pharmacokinetic parameter: Cmax | Day 1 pre-dose and 0.75, 1.25, 2.25, 4.25 6.25, 8.25 and 12.25 hours post-dose and on Days 2 and 3 at 24.25, 32.25 and 48.25 hours
  Apparent maximum plasma concentration (will be directly read from the measured concentration-time profile)
Pharmacokinetic parameter: tmax | Day 1 pre-dose and 0.75, 1.25, 2.25, 4.25 6.25, 8.25 and 12.25 hours post-dose and on Days 2 and 3 at 24.25, 32.25 and 48.25 hours
  Time to reach the apparent maximum plasma concentration (will be directly obtained from the blood sampling time as time from administration to the time of first occurrence of Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- DecisionLine Clinical Research Corporation, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No